CLINICAL TRIAL: NCT06328725
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase 1/2 Trial to Evaluate the Efficacy and Safety of EN001 in Patients With Duchenne Muscular Dystrophy
Brief Title: Evaluate the Efficacy and Safety of EN001 in Patients With Duchenne Muscular Dystrophy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ENCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN001_POWER
Record Dates: First submitted 2024-02-19; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: <Phase 1 Clinical Trial> A total of 6-12 participants (3-6 participants per cohort).
  <Phase 2 Clinical Trial> A total of 76 participants (a minimum of 30 participants per group, considering a dropout rate of 20%, resulting in 38 participants per group).
Who Masked: Participant, Investigator
Masking Description: The investigational drug for the clinical trial of the following cohort or group will be administered intravenously (IV) three times at 6-week intervals.
  <Phase 1 Clinical Trial> Cohort 1: EN001 5.0x10^5 cells/kg / Cohort 2: EN001 2.5x10^6 cells/kg
  <Phase 2 Clinical Trial> Experimental Group: Recommended Phase 2 Dose (RP2D) for EN001 / Control Group: Placebo for EN001
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 - Cohort 1 (Active Comparator): EN001 5.0x10^5 cells/kg
  Interventions: Drug: EN001
- Phase 1 - Cohort 2 (Active Comparator): EN001 2.5x10^6 cells/kg
  Interventions: Drug: EN001
- Phase 2 - Experimental Group (Placebo Comparator): The recommended phase 2 dose (RP2D) of EN001
  Interventions: Drug: EN001
- Phase 2 - Control Group (Placebo Comparator): EN001 placebo
  Interventions: Drug: EN001

INTERVENTIONS:
Drug: EN001 — Phase 1
  * Cohort 1: EN001 5.0x10^5 cells/kg administered intravenously (IV) 3 times at 6 week intervals.
  * Cohort 2: EN001 2.5x10^6 cells/kg administered intravenously (IV) 3 times at 6 week intervals.
  Phase 2
  * Experimental Group: The recommended phase 2 dose (RP2D) of EN001 is administered intravenously (IV) three times at six-week intervals.
  * Control Group: EN001 placebo is administered intravenously (IV) three times at six-week intervals.
  Other Names: EN001(allogenic early-passage mesenchymal stem cells derived from Wharton's jelly (WJ-MSCs) )

SUMMARY:
A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase 1/2 Trial to Evaluate the Efficacy and Safety of EN001 in Patients with Duchenne Muscular Dystrophy

DETAILED DESCRIPTION:
This clinical trial is a multi-center study conducted in two phases: Phase 1 and Phase 2. Phase 1 follows a 3+3 dose-escalation design to assess the safety, efficacy, and tolerability of EN001, an investigational product. Phase 2 evaluates the efficacy and safety of EN001 at the recommended phase 2 dose (RP2D), as determined in Phase 1, compared to a placebo.

Phase 1 is designed using the traditional 3+3 dose-escalation method to determine the maximum tolerated dose (MTD) and establish the RP2D. Dose escalation continues until the MTD is identified, which must be within the maximum planned dose (MPD) of 2.5 x 10^6 cells/kg (Cohort 2) or lower. The MTD is defined as the highest dose at which the incidence rate of dose-limiting toxicity (DLT) is less than 33%. To determine the MTD, 3-6 subjects are enrolled in each dose cohort. They receive EN001 every 6 weeks for 3 cycles, with DLTs evaluated up to the 2-week time point (Visit 7).

The Safety Review Committee (SRC) consists of the coordinating Investigator, the responsible trial monitor for subjects enrolled in cohorts requiring safety review, and the sponsor. These members participate as committee members. At the conclusion of each cohort-defined as the endpoint of the DLT assessment for the last subject in that cohort-they comprehensively review the safety data for EN001. The committee makes decisions related to dose adjustments, whether to increase or decrease the dose, and ultimately determines the RP2D.

Phase 2 clinical trials are randomized, double-blind, placebo-controlled clinical trials.

In phase 2, eligible subjects will be randomly assigned to the test group (recommended phase 2 dose (RP2D) of EN001) or the control group (placebo of EN001) in a 1:1 ratio. Efficacy and safety will be evaluated up to 48 weeks after EN001 administration compared to placebo.

In addition, test subjects participating in phase 1 and phase 2 will be followed up for safety and effectiveness for 5 years from the time of EN001 administration according to the long-term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged between 6 and 11 years at the time of providing written consent.
2. Individuals exhibiting phenotypic signs of Duchenne Muscular Dystrophy (DMD), such as lower limb muscle weakness, a duck walk, or Gower's sign, and who are diagnosed with DMD following confirmation of a dystrophin gene mutation through genetic testing.
3. Participants who meet the Time to Stand Test (TTSTAND) criteria without the use of assistive devices or help from others during screening and baseline assessments:

   * Phase 1: Capable of completing the TTSTAND evaluation.
   * Phase 2: TTSTAND time of 10 seconds or less.
4. Participants with a 6-Minute Walk Test (6MWT) result of 75 meters or more at screening and baseline.
5. Individuals who meet the following laboratory test criteria at the time of screening and baseline:

   * Hemoglobin ≥10 g/dL
   * Platelet ≥50,000/μL
   * Serum albumin ≥2.5 g/dL
   * Gamma glutamyl transferase (γ-GT) and total bilirubin ≤ upper limit of normal (ULN)
   * Serum creatinine ≤ 1.5 x ULN
6. Participants who have been on a stable dose of glucocorticoids for at least 12 weeks prior to screening, with treatment maintained. Dosage adjustments for body weight changes are allowed.
7. Individuals who, along with their representatives when applicable, have voluntarily agreed in writing to participate in this clinical trial.

Exclusion Criteria:

1. Individuals with confirmed comorbidities at the time of screening:

   * Left ventricular ejection fraction (LVEF) below 50%, as determined by echocardiography
   * Percent predicted forced vital capacity (FVC%) less than 35%
   * Positive for Hepatitis B surface antigen (HBsAg). However, individuals undergoing interferon or antiviral treatment can register
   * Positive for Hepatitis C virus antibody (HCV Ab). Registration is possible if the HCV ribonucleic acid (RNA) test result is negative
   * Positive for Human immunodeficiency virus (HIV) antibody
   * Comorbidities that are uncontrollable or require treatment that could affect the safety and efficacy evaluation of this clinical trial, based on the investigator's judgment
2. Individuals with confirmed treatment history at the time of screening:

   * Administration of cell therapy or gene therapy throughout life
   * Administer antisense oligonucleotide (e.g., exon skipping treatment) or stop- codon readthrough treatment (e.g., aminoglycoside, ataluren) within 24 weeks before screening.
   * Administration of the following medications within 12 weeks before screening: Idebenone, Resveratrol, Adenosine triphosphate
   * Administration of the following medications within 12 weeks before screening. However, registration is possible if the drug is being administered at a stable dose for at least 12 weeks before screening and the dose is expected to remain unchanged during the clinical trial period. Angiotensin-converting enzyme (ACE) inhibitor Angiotensin II receptor blocker (ARB) Beta-blocker Aldosterone antagonist Ivabradine Sacubitril Growth hormone Anabolic steroids
   * Major surgery within 12 weeks before screening or expected major surgery during the clinical trial period.
   * Use of other investigational products (or medical devices) within 4 weeks before screening.
   * Use of systemic immunosuppressants other than systemic glucocorticoids.
3. Individuals requiring mechanical ventilation during the day.
4. Persons with hypersensitivity to the components of the clinical investigational products.
5. Individuals unwilling to use appropriate contraception from the date of written consent to the termination visit:

   * Appropriate contraceptive methods are as follows, and use more than one method.

     * The use of hormonal contraceptives by the partner
     * Implantation of an intrauterine device or system in your partner
     * Sterilization or surgical procedures for you or your partner
6. Others who, in the investigator's discretion, are not willing or able to comply with the clinical trial procedures.

Ages: 6 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
<Phase 1> Adverse drug reactions related to dose limiting toxicity (DLT) | Up to 14 weeks
  Present the frequency and percentage of dose-limiting toxicity (DLT) occurrence across dose cohorts, along with detailed information on the types of DLTs.
<Phase 1> Adverse drug reactions related to discontinuation of clinical trial drug administration | Up to 14 weeks
  Present the frequency and percentage of dose-limiting toxicity (DLT) occurrence across dose cohorts, along with detailed information on the types of DLTs.
<Phase 2> Change in time to stand test (TTSTAND) | At 48 weeks compared to baseline (Visit 2)
  Present the changes in time to stand test (TTSTAND) at the 48-week time point compared to baseline (Visit 2). Provide the subject count, mean, standard deviation, median, minimum, and maximum for the change in each treatment group. Analyze the change as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline TTSTAND values and age as fixed effects in the analysis.

SECONDARY OUTCOMES:
<Phase 1> Time to stand test (TTSTAND) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> TTSTAND velocity (1/TTSTAND) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> Time to run/walk 10 meters test (TTRW) change amount | At 6, 12, 18, 24, 36,, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> TTRW velocity (1/TTRW) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> North Star Ambulatory Assessment (NSAA) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> Time to climb 4 steps test (TTCLIMB) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> TTCLIMB velocity (1/TTCLIMB) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> 6-minute walk test (6MWT) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> Changes amount in muscle strength by region | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  The changes in shoulder abduction, elbow flexion/extension, knee flexion/extension, and handgrip are evaluated using hand-held myometry. (Unit: lbs)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> Changes amount in parameters related to pulmonary function | At 12, 24, and 48 weeks compared to baseline (Visit 2)
  Through spirometry testing, % predicted forced vital capacity (FVC%), forced vital capacity (FVC, unit L), forced expiratory volume in one second (FEV1), peak expiratory flow rate (PEFR), maximal inspiratory pressure (MIP), maximal expiratory pressure (MEP).
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> Changes amount in parameters related to cardiac function | At 48 weeks compared to screening (Visit 1)
  Through echocardiography, changes in left ventricular ejection fraction (LVEF), fractional shortening (FS), and left ventricular end-diastolic diameter (LVEDd) are evaluated.
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 1> Change rate of creatine kinase (CK) at each visit after administration of investigational product compared to baseline (Visit 2) | From baseline
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
<Phase 2> Time to stand test (TTSTAND) change amount | At 6, 12, 18, 24, and 36 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> TTSTAND velocity (1/TTSTAND) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Time to run/walk 10 meters test (TTRW) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> TTRW velocity (1/TTRW) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> North Star Ambulatory Assessment (NSAA) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Time to climb 4 steps test (TTCLIMB) change | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> TTCLIMB velocity (1/TTCLIMB) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> 6-minute walk test (6MWT) change amount | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Changes amount in muscle strength by region | At 6, 12, 18, 24, 36, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Changes amount and rate of change in whole thigh muscle volume and index assessed by MRI | At 48 weeks compared to screening (Visit 1)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Changes amount in parameters related to pulmonary function | At 12, 24, and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Changes amount in parameters related to cardiac function | At 48 weeks compared to screening (Visit 1)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Change rate of creatine kinase (CK) at each visit after administration of investigational product compared to baseline (Visit 2) | From baseline
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Pediatric Outcomes Data Collection Instrument (PODCI) item score and total score change | At 24 and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 2> Pediatric Quality of Life inventory™ (PedsQL™) item scores and total score change | At 24 and 48 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for changes at each time point and for each dosage group. Analyze the change (or percentage change) as the dependent variable using a repeated measures mixed model (MMRM) with treatment group, visit (6, 12, 18, 24, 36, 48 weeks), and the interaction between treatment group and visit as factors. Include baseline (or screening) values of each assessment variable, age, and a stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as fixed effects in the analysis. However, for variables related to TTSTAND, do not include the stratification factor (TTSTAND ≤ 8 seconds / > 8 seconds) as a fixed effect.
<Phase 1> Adverse Event | Up to 48weeks. However, adverse drug reactions that persist at the end of the clinical trial will be followed up until the possible adverse reactions are resolved or it is determined that further follow-up is not meaningful.
  After the application of the investigational medicinal product in the clinical trial, provide the number of subjects, incidence rate, and number of occurrences for adverse events, drug-related adverse events, serious adverse events, serious drug-related adverse events, adverse events related to discontinuation of the investigational medicinal product, drug-related adverse events related to discontinuation of the investigational medicinal product, and injection-related adverse events, categorized by dosage group. Additionally, code the occurrences by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA), and present the number of subjects, incidence rate, and number of occurrences for each dosage group according to SOC and PT.
<Phase 1> Laboratory examination | Up to 48weeks. At Baseline and Week 4, tests are conducted before and within 4 hours after administration of the investigational drug, and PT INR and aPTT are performed only at the screening visit.
  Number of participants with clinically significant abnormalities in Laboratory parameters after EN001 administration.
  Hematological tests, Blood chemical tests, Blood coagulation test, Urine test, Serum virus test
  It is conducted through blood and urine collection, and the PI checks whether the test results are normal, abnormal, and clinically significant.
<Phase 1> Vital sign | Up to 48weeks.
  Number of participants with clinically significant abnomalities in vital signs after EN001 administration.
  Vital Signs include blood pressure (mmHg), pulse (times/minute), respiratory rate (times/minute), and body temperature (℃) and will be assessed.
  For changes at each time point within each dosage group, present continuous variables with subject count, mean, standard deviation, median, minimum, and maximum. For categorical variables, provide frequency and percentage.
<Phase 2> Adverse Event | Up to 48weeks. However, adverse drug reactions that persist at the end of the clinical trial will be followed up until the possible adverse reactions are resolved or it is determined that further follow-up is not meaningful.
  After the administration of the investigational product in the clinical trial, provide the number of subjects, incidence rate, and number of occurrences for adverse events, drug-related adverse events, serious adverse events, serious drug-related adverse events, adverse events related to discontinuation of the investigational product, drug-related adverse events related to discontinuation of the investigational product, and injection-related adverse events, categorized by treatment group. Additionally, code the occurrences by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA), and present the number of subjects, incidence rate, and number of occurrences for each treatment group according to SOC and PT.
<Phase 2> Laboratory examination | Up to 48weeks. At Baseline and Week 4, tests are conducted before and within 4 hours after administration of the investigational drug, and PT INR and aPTT are performed only at the screening visit.
  Number of participants with clinically significant abnormalities in Laboratory parameters after EN001 administration.
  Hematological tests, Blood chemical tests, Blood coagulation test, Urine test, Serum virus test
  It is conducted through blood and urine collection, and the PI checks whether the test results are normal, abnormal, and clinically significant.
<Phase 2> Vital sign | Up to 48weeks.
  Number of participants with clinically significant abnomalities in vital signs after EN001 administration.
  Vital Signs include blood pressure (mmHg), pulse (times/minute), respiratory rate (times/minute), and body temperature (℃) and will be assessed.
  For changes at each time point within each treatment group, present continuous variables with subject count, mean, standard deviation, median, minimum, and maximum. For categorical variables, provide frequency and percentage.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul